CLINICAL TRIAL: NCT00885144
Title: Differential Acceptability of New Lipid Based Nutrient Supplement (LNS) Formulations for Prevention of Moderate Malnutrition
Brief Title: Trial on the Acceptability of Modified Lipid Based Nutrient Supplements Among Malawian Infants
Acronym: iLiNS-ACCEPT-M
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tampere University (Other)
Collaborators: Kamuzu University of Health Sciences (Other); University of California, Davis (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Per Ashorn / Professor of International Health, University of Tampere
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: iLiNS-ACCEPT-M
Record Dates: First submitted 2009-04-20; First posted 2009-04-21 (Estimated); Last update posted 2009-06-24 (Estimated); Status verified 2009-06

CONDITIONS: Malnutrition
Keywords: Stunting; Growth failure; Malnutrition; Lipid based nutrient supplement; LNS; Prevention; Malawi; Sub-Saharan Africa; Dietary supplementation
MeSH Terms: conditions — Malnutrition; Growth Disorders; Failure to Thrive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Nutributter — Test dose of "standard" supplementary lipid based nutrient supplement (LNS). 15 grams of Nutributter will be mixed with 30 g of maize porridge and fed to the child over a maximum of 15 minute period, under direct observation.
Dietary Supplement: LNS-20gM — Test dose of modified LNS-20gM supplementary lipid based nutrient supplement (LNS). 15 grams of LNS-20gM will be mixed with 30 g of maize porridge and fed to the child over a maximum of 15 minute period, under direct observation.
Dietary Supplement: LNS-20gNoM — Test dose of modified LNS-20gNoM (milk free) supplementary lipid based nutrient supplement (LNS). 15 grams of LNS-20gNoM will be mixed with 30 g of maize porridge and fed to the child over a maximum of 15 minute period, under direct observation.
Dietary Supplement: LNS-10gM — Test dose of modified LNS-10gM supplementary lipid based nutrient supplement (LNS). 15 grams of LNS-10gM will be mixed with 30 g of maize porridge and fed to the child over a maximum of 15 minute period, under direct observation.

SUMMARY:
The use of lipid-based nutrients (LNS), such as Nutributter or fortified spread (FS), have been associated with improved growth and development outcomes among infants in Ghana and Malawi. The investigators' study group has developed modified versions of such supplements that theoretically will supplement infants diets better and with lower cost. As a preparation for larger efficacy trials, the investigators now aim to test the acceptability of these supplements among Malawian infants and their guardians. The trial hypothesis is that the infants will consume on average at least 50% of an offered dose that consists of LNS mixed with maize porridge.

DETAILED DESCRIPTION:
In the first phase, 18 infants meeting set criteria are randomised into receiving three test meals with novel LNS preparations over a three-day period. The meals will consists of the following, each given on one day and in a random order: 1) 7.5 g of LNS-10gM mixed in 30 g maize-soy porridge, 2) 15 g of LNS-20gM mixed in 30 g maize-soy porridge, 3) 15 g of LNS-20gNoM mixed in 30 g maize-soy porridge. As a run in procedure, each participant will undergo a test feeding session with one of the the test foods on the day before the actual test-feeding period. As a positive control, each participant will undergo test feeding session with standard Nutributter (NB) on the day after the actual test-feeding period.

In the second phase a set of 48 infants are randomised into 3 groups receiving the following food supplements for a period of 2 weeks: 1) 10 g/day of milk-containing, very concentrated LNS (LNS-10gM), 2) 20 g/day of milk-containing, concentrated LNS (LNS-20gM), 3) 20 g/day of milk-free, concentrated LNS (LNS-20 g NoM)

Outcomes measures in the first phase will be assessed through safety reports and quantities of test food consumed by the child and a hedonic scale of acceptability by the mothers of the children. The second phase will be assessed with qualitative outcomes, from data obtained from focus group discussions with the guardians of the infants consuming the test foods.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent from at least one guardian
* Age 7.50 months to 11.49 months
* Currently breastfeeding
* Consuming complementary feeds at least 30 days prior to enrollment
* Availability during the period of the study

Exclusion Criteria:

* Weight for length Z score (WFH) ≤ -2.0 using WHO growth reference standards or the -presence of oedema
* Severe systemic illness warranting hospital referral
* History of allergy towards peanut
* History of anaphylaxis or serious allergic reaction to any substance, requiring emergency medical care
* Congenital malformation such as cleft palate which may interfere with food intake
* Concurrent participation in any other clinical trial

Ages: 8 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2009-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Mean amount (in grammes) of test food consumed | within 15 minutes of test feeding

SECONDARY OUTCOMES:
Mean time taken to consume the intervention dose | 15 minutes after test feeding
Mean rating by the guardians (on a hedonic, 5 point scale) | 15 minutes after test feeding
Overall guardian feedback after a two week supplementation period (qualitative analysis of focus group discussions) | Once, when the children have completed a two-week supplementary feeding period

CONTACTS AND LOCATIONS:
Overall Officials: Per Ashorn, MD, PhD, Principal Investigator — Tampere University; Kenneth Maleta, MBBS, PhD, Principal Investigator — Kamuzu University of Health Sciences
Locations (1):
- University of Malawi, College of Medicine, Mangochi, Malawi

REFERENCES:
- See also: College of Medicine homepage — http://www.medcol.mw/